CLINICAL TRIAL: NCT02744807
Title: Prevalence of Chronic Endometritis in Severe Intrauterine Adhesions and Role of Chronic Endometritis in Postoperative Recurrence of Severe Intrauterine
Brief Title: Role of Chronic Endometritis in Postoperative Recurrence of Severe Intrauterine Adhesions
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yuqing Chen, Deputy chief physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 2013B021800237
Record Dates: First submitted 2016-04-10; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Intrauterine Adhesions; Chronic Endometritis
Keywords: intrauterine adhesions; Chronic endometritis; infections; Hysteroscopy
MeSH Terms: conditions — Gynatresia; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrium
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- non-Chronic endometritis: patients with intrauterine adhesion only
- Chronic endometritis: patients with intrauterine adhesion as well as Chronic endometritis
  Interventions: Other: Chronic endometritis

INTERVENTIONS:
Other: Chronic endometritis — with or without Chronic endometritis
  Groups: Chronic endometritis

SUMMARY:
This study is to evaluate the prevalence of chronic endometritis (CE) in women with severe intrauterine adhesions and compare recurrence of adhesion in women with and without CE.

DETAILED DESCRIPTION:
Chronic endometritis (CE) is a persistent in endometrium that is characterized by the presence of plasma cells. Recently, there has been increasing interest in the role of CE in recurrent pregnancy loss (RPL). One of the most common uterine abnormalities for RPL is Intrauterine adhesion (IUA).Intrauterine adhesion, also known as Asherman's syndrome, is the partial or complete occlusion of the uterine cavity as a result of endometrium damage. Most intrauterine adhesions patients manifest amenorrhea, reduced menstrual pattern, infertility, and intrauterine growth restriction, which seriously affect their reproductive health.It is well established that the formation of IUA likely involves hypoxia, reduced neovascularization, and altered expression of adhesion-associated cytokines, but the exact mechanisms are not well understood. Although excessive curettage is considered the primary cause, intrauterine adhesion is known to be associated with diverse non-traumatic factors, such as postabortal sepsis, puerperal sepsis and infections. It is therefore possible to hypothesize that Intrauterine adhesion may be related to chronic endometritis. To the best of researchers knowledge,there have been no reports investigating this relationship. The aim of this study was to clarify the hypothesis by evaluating the prevalence of chronic endometritis (CE) in women with severe intrauterine adhesions and compare recurrence of adhesion in women with and without chronic endometritis (CE).

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative adhesion score was ≥5
* The prior menstrual cycle was regular, and the sex hormone was normal
* with informed consent
* absence of other uterine abnormality at transvaginal ultrasound
* There were no severe systemic diseases, and no contradictions to aspirin, estrogen and surgery.

Exclusion Criteria:

* Pre-operative adhesion score was <5
* Prior menstrual cycle was irregular and sex hormone was abnormal, or patients had endocrine factors that caused amenorrhea, menstrual reduction and infertility
* other uterine abnormality at transvaginal ultrasound
* without informed consent
* Patients had contradictions to estrogen and aspirin such as cancers (breast cancer and endometrial cancer), thrombotic diseases, allergy to antipyretic analgesics, severe liver injury, hypoprothrombinemia, vitamin K deficiency, hemophilia, thrombocytopenia, gastric or duodenal ulcer and asthma
* refuse Endometrial biopsy
* Vaginal discharge abnormal, or Suspected vaginitis or pelvic inflammatory disease, or using antibiotics.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 125 patients who received hysteroscopy in the Department of Obstetrics and Gynecology of the First Affiliated Hospital of Sun Yat-sen University and were diagnosed with moderate to severe Intrauterine adhesion according to the criteria of American Fertility Society (AFS) were recruited into present study.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants With recurrence of adhesion in women with and without Chronic endometritis | 1 year
  Second-look hysteroscopy was carried out in the early proliferative phase, 1 to 3 months after the initial operation.After assessment of the extent and severity of any reformed adhesions, hysteroscopic adhesiolysis was also carried out at the time of the second-look procedure, if adhesions had recurred.

SECONDARY OUTCOMES:
Reduction of American Fertility Society adhesion score at Second-look hysteroscopy between women with and without Chronic endometritis | 1 year
  The severity and extent of intrauterine adhesions were scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version) [7]. A score of 1-4 was considered to represent mild adhesions, a score of 5-8 was considered to represent moderate adhesions and a score of 9-12 represented severe adhesions.
Number of patients diagnosed with Chronic endometritis at hysteroscopy | 1 year
  Chronic endometritis signs at hysteroscopy included [1] pedunculated and vascularized micro-polyps (<1 mm), most frequently found near the endocervical area (2); and [2] the presence of areas of hyperemic endometrium flushed with a white central point, localized or scattered throughout the cavity, referred to as "strawberry aspect".
Number of patients with Chronic endometritis confirmed by histology | 1 year
  Endometrial samples were fixed in neutral formalin and later embedded in paraffin for histological analysis. Five-micrometer sections were stained with hematoxilin-eosin. Histological diagnosis of Chronic endometritis: Attention was paid to the following features: superficial stromal edema, increased stromal density, pleomorphic stromal inflammatory infiltrate dominated by lymphocytes and plasma cells.

CONTACTS AND LOCATIONS:
Overall Officials: chen yu qing, Deputy chief, Principal Investigator — The First Affiliated Hospital of SunYetSen University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] McQueen DB, Perfetto CO, Hazard FK, Lathi RB. Pregnancy outcomes in women with chronic endometritis and recurrent pregnancy loss. Fertil Steril. 2015 Oct;104(4):927-931. doi: 10.1016/j.fertnstert.2015.06.044. Epub 2015 Jul 21. PMID 26207958
- [Derived] Liu L, Yang H, Guo Y, Yang G, Chen Y. The impact of chronic endometritis on endometrial fibrosis and reproductive prognosis in patients with moderate and severe intrauterine adhesions: a prospective cohort study. Fertil Steril. 2019 May;111(5):1002-1010.e2. doi: 10.1016/j.fertnstert.2019.01.006. Epub 2019 Mar 25. PMID 30922643
- [Derived] Chen Y, Liu L, Luo Y, Chen M, Huan Y, Fang R. Prevalence and Impact of Chronic Endometritis in Patients With Intrauterine Adhesions: A Prospective Cohort Study. J Minim Invasive Gynecol. 2017 Jan 1;24(1):74-79. doi: 10.1016/j.jmig.2016.09.022. Epub 2016 Oct 20. PMID 27773811